CLINICAL TRIAL: NCT00596882
Title: Message Priming and Enrollment in, and Response to, a Smoking Cessation Program: A Pilot Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Pennsylvania Department of Health (Other Government); Pfizer (Industry)
Responsible Party: Robert Schnoll, Ph.D., University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 806910
Record Dates: First submitted 2008-01-08; First posted 2008-01-17 (Estimated); Last update posted 2009-12-02 (Estimated); Status verified 2009-12

CONDITIONS: Smoking Cessation
Keywords: smoking cessation; nicotine dependence; message prime; recruitment
MeSH Terms: conditions — Smoking Cessation; Tobacco Use Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Other): Threat only message. Participants hear information about the negative health consequences of smoking
  Interventions: Other: Message Prime
- 2 (Other): Genetic threat + threat. Participants will bear infomration about genetic influences of smoking in additon to the negative health consequences of smoking.
  Interventions: Other: Message Prime

INTERVENTIONS:
Other: Message Prime — Participants will be randomized to genetic prime messages or threat only message at the time of the intial telephone screen. Following phone screen, all eligibleparticipants will receive 13 weeks of Chantix with smoking cessation counseling.
Other: Message Prime — Particpants will be randomized into 1 of 2 groups. 1 group will recieve a message detailing the negative helaht consequenes of smoking and the other group will receive this information along with information about the genetic incluences on smoking behavior.

SUMMARY:
The proposed study has been designed to examine the effect of a message that primes genetic susceptibility on actual enrollment in a smoking cessation program, actual response to smoking cessation treatment, and potential moderators and mediators of this effect.

DETAILED DESCRIPTION:
Despite available behavioral and pharmacological interventions to treat nicotine dependence, most smokers do not utilize these interventions. As such, the vast majority of smokers do not capitalize on potentially effective nicotine dependence treatments. The way in which health risk information is presented may influence interest in a smoking cessation program. In a series of preliminary studies, individuals provided with messages that primed the role of genetic variation in susceptibility to addiction to smoking exhibited positive consequences on intentions to quit (Cappella, Lerman, Romantan, & Baruh, 2005). The proposed study has been designed to examine the effect of a message that primes genetic susceptibility on actual enrollment in a smoking cessation program, actual response to smoking cessation treatment, and potential moderators and mediators of this effect. The results of this pilot study may provide preliminary data for a larger trial and have implications for designing interventions to promote utilization of effective treatments for nicotine dependence among smokers.

ELIGIBILITY:
Eligible participants will be 100 male & female smokers aged 18-65, who smoke ≥ 10 cigarettes/day & who plan to live in the area for the next 6-months.

Key Exclusion Criteria Smoking Behavior

1.Use of chewing tobacco or snuff 2.Current enrollment or plans to enroll in another smoking cessation program in the next 6 months 3.Plan to use other nicotine substitutes or smoking cessation treatments in the next 6 months Alcohol/Drug Exclusion Criteria

1. History of substance abuse and/or currently receiving treatment for substance abuse
2. Current alcohol consumption that exceeds >25 standard drinks/week

Medication Exclusion Criteria

1. Current use or recent discontinuation (within last 14-days) of the following medications:

   1. Any form of smoking cessation medication
   2. Any form of anti-psychotic medications that includes:

      •antipsychotics,

      •atypical antipsychotics,

      •mood-stabilizers,

      •anti-depressants (tricyclics, SSRI's, MAOI's),

      •anti-panic agents,

      •anti-obsessive agents,

      •anti-anxiety agents, and
      * stimulants (e.g., Provigil, Ritalin).
   3. Medication for chronic pain
   4. Anti-coagulants
   5. Any heart medications
   6. Daily medication for asthma

Medical Exclusion Criteria

1. Women who are pregnant, planning a pregnancy, or lactating.
2. History or current diagnosis of psychosis, major depression or bipolar disorder, schizophrenia, or any Axis 1 disorder.
3. Serious/unstable disease within the past 6 months (e.g., cancer [but melanoma], heart disease, HIV).
4. History of epilepsy or a seizure disorder.
5. History or current diagnosis (last 6-months) of abnormal rhythms and/or tachycardia (>100 beats/minute); history or current diagnosis of COPD, cardiovascular disease (stroke, angina, coronary heart disease), heart attack in the last 6 months, uncontrolled hypertension (SBP>150 or DBP>90).
6. History of kidney and/or liver failure (including transplant).

General Exclusion

1. Any medical condition or concomitant medication that could compromise participant safety or treatment, as determined by the Principal Investigator and/or Study Physician.
2. Inability to provide informed consent or complete any of the study tasks as determined by the Principal Investigator and/or Study Physician.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2008-02; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
The primary outcome variables are:(1)Attendance to the intake evaluation & enrollment in the smoking cessation program; (2)7-day point prevalence abstinence(3)Self-reported cigarette consumption | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Robert Schnoll, Ph.D., Principal Investigator — University of Pennsylvania
Locations (1):
- Transdisciplinary Tobacco Use Research Center, Philadelphia, Pennsylvania, United States